CLINICAL TRIAL: NCT03612141
Title: Extern Validation of a Predictive Score of Brain Death in Patients With Severe Stroke and Unfavourable Prognosis Identified by Organ Procurement and Transplant Coordinations
Brief Title: Extern Validation of a Predictive Score of Brain Death in Severe Stroke (DIAPASON1)
Acronym: DIAPASON1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02087-48
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Stroke
Keywords: Severe stroke; Brain Death; organ donation
MeSH Terms: conditions — Stroke; Brain Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is currently a shortage of organ in France, for patients with chronic diseases who are on the waiting list for an organ. The first source of organ donor in France is patients with brain death. 58% of patients in brain death are patients with a severe stroke ( ischemic or hemorrhagic). In order to identify which patient with a severe stroke and with unfavorable prognosis who can evolve to brain death, we have conducted a retrospective study in Lorrain, in France, and we have built a predictive score of brain death in these patients. It is important to validate this predictive score in a prospective study on a greater scale than the first study.

DETAILED DESCRIPTION:
Main objective :

External validation of a brain death evolution predictive score GRAHAL65 (initial Glasgow score ≤6, systolic blood pressure >150 mmHg, past history of alcohol abuse, herniation, hydrocephalus, and stroke volume>65 ml) for patients with severe stroke and withhold therapy built.

Secondary objectives :

Identification of other clinical and paraclinical predictive factors of brain death evolution:

* Age,sex,
* Temperature and glycemia
* Rostro-caudal abolition of brainstem reflexes
* Other cardiovascular risk factors (hypertension, diabetes, atrial fibrillation, dyslipidemia,)
* Antiplatelet therapy, anticoagulant treatment,
* Intravenous thrombolytic therapy or thrombectomy
* Type of stroke
* Infarct location
* Type of brain herniation

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years and over.
* Patient with a sever stroke less than 48 hours diagnosed by brain imaging magnetic resonance imaging or computed tomography (including cerebral infarction, intra-parenchymal hemorrhage and subarachnoid haemorrhage
* Patient with Glasgow Scale score <8 Engaged vital prognosis
* Absence of therapeutic resources
* Decision of resuscitation measures to protect the organs in the purpose organ donation after brain death

Exclusion Criteria:

* Pregnant woman
* Patient with recent traumatic brain injuries (subdural hematoma, extradural hematoma and contusions)
* Obvious contraindication of organ donation excluding the patient from organ protection measures in intensive care unit (expression of patient opposition, HIV infection, active tuberculosis, spongiform encephalopathy,
* human growth hormones treatment origin, rabies, active cancer)
* Opposition of family member of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be included in this study will be
  * Patients with a severe stroke admitted in a stroke unit or a intensive care unit
  * With a engaged vital prognosis ( life threatened pateint)
  * With non opposition to organ donation
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Brain death | 5 days
  Brain death defined confirmed by the mandatory criteria of the current French legislation for organ procurement including in the absence of confounding factors such as sedation, deep hypothermia, severe metabolic disorders):
  * clinical assessment (absence of consciousness (Glasgow score =3), absence of spontaneous respiration absence of brain stem reflexes)
  * paraclinical assessment: two flat and areactive electroencephalography recordings or cerebral angiography/cerebral CT scanshowing no cerebral circulation

CONTACTS AND LOCATIONS:
Locations (25):
- France (25):
  - CH d'Auxerre, Auxerre
  - Hôpital Nord Franche, Belfort
  - CHU Besançon, Besançon
  - CH de Charleville-Mézières, Charleville-Mézières
  - CH de Chalons-en-Champagne, Châlons-en-Champagne
  - CH de Colmar, Colmar
  - Ch de Compiègne, Compiègne
  - CHU de Dijon, Dijon
  - CH Epinal, Épinal
  - CH de Haguenau, Haguenau
  - CH de Laon, Laon
  - Lons Le Saunier, Lons-le-Saunier
  - CH de Macon, Mâcon
  - CHR Metz-Thionville, Metz
  - CH de Mulhouse, Mulhouse
  - CHRU de Nancy, Nancy
  - CH Nevers, Nevers
  - CHU de Reims, Reims
  - CH de Saint-Quentin, Saint-Quentin
  - CH Sarreguemines, Sarreguemines
  - CH de saverne, Saverne
  - CHRU de Strasbourg, Strasbourg
  - CH Troyes, Troyes
  - CH Verdun, Verdun
  - CH de Vesoul, Vesoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Humbertjean L, Mione G, Fay R, Durin L, Planel S, Lacour JC, Enea AM, Richard S. Predictive factors of brain death in severe stroke patients identified by organ procurement and transplant coordination in Lorrain, France. Transpl Int. 2016 Mar;29(3):299-306. doi: 10.1111/tri.12695. PMID 26402792